CLINICAL TRIAL: NCT03302221
Title: Regional Haemodynamic Changes in Radial Artery Assessment With Continuous Pulsed-wave Doppler Ultrasound in Patients Undergoing Video-assisted Thoracic Surgery With Different Kinds of Anaesthesia Management
Brief Title: Regional Haemodynamic Changes in Radial Artery Assessment With Continuous Pulsed-wave Doppler Ultrasound
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Associate proffesor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170711-01
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Doppler Ultrasonography Assessed Vascular Changes
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group control (Other): In the control group, local anaesthesia at the incision was induced by 0.5% ropivacaine by the surgeon just before the surgery.
  Interventions: Drug: 0.5% ropivacaine local anaesthesia
- Paravertebral Block Group (Experimental): In Group Paravertebral Block, patients received standardized general anaesthesia supplemented by paravertebral Block. The USG approach for TPVB was used with the patient in the lateral position at the T4-T6 level according to the incision protocol in our centre.
  Interventions: Drug: 0.5% ropivacaine paravertebral block
- Epidural Block Group (Experimental): The investigators designed a study to assess whether there were any blood flow indexes change during induction with doppler ultrasonography ;general anesthesia combined with epidural block
  Interventions: Drug: 0.25% ropivacaine epidural block

INTERVENTIONS:
Drug: 0.5% ropivacaine paravertebral block — The investigators designed a study to assess whether there were any blood flow indexes change during induction with doppler ultrasonography after 0.5% ropivacaine paravertebral block
  Arms: Paravertebral Block Group
Drug: 0.25% ropivacaine epidural block — A 4-5 ml bolus of 0.25% ropivacaine was administered 1 h after the initiation of TEB.
  Arms: Epidural Block Group
Drug: 0.5% ropivacaine local anaesthesia — local anaesthesia at the incision was induced by 0.5% ropivacaine by the surgeon just before the surgery.
  Arms: Group control

SUMMARY:
The objective of the trial was to evaluate velocity-associated parameters of pulsed-wave Doppler ultrasound at induction, discharge from the post-anaesthesia care unit and during inspiratory cough in addition to the consumption of phenylephrine during the operation in patients undergoing video-assisted thoracic surgery with three types of anaesthesia management.

DETAILED DESCRIPTION:
The objective of the trial was to evaluate velocity-associated parameters of pulsed-wave Doppler ultrasound at induction, discharge from the post-anaesthesia care unit and during inspiratory cough in addition to the consumption of phenylephrine during the operation in patients undergoing video-assisted thoracic surgery with three types of anaesthesia management. The patients in this trial were visited during the entire operation and just before leaving the post-anaesthesia care unit. Velocity-associated data related to pulsed-wave Doppler ultrasound and the consumption of phenylephrine were collected.

ELIGIBILITY:
Inclusion Criteria:

1. ethnic Chinese;
2. age, 18 to 65 years old;
3. American Society of Anaesthesiologists (ASA) physical status I or II;
4. required VATS for lung surgery and one lung ventilation .

Exclusion Criteria:

body mass index exceeding 30 kg/m2; Patients with a history of hypertension, diabetes mellitus or arteriosclerosis; and any allergy to drugs used in the study.

Patients with arrhythmias or implanted cardiac pacemakers were excluded. Patients with diseases of the central or peripheral nervous system were excluded.

Patients taking medications affecting the autonomic nervous system, such as b-blockers and calcium channel blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-08-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
The Change of end-diastolic velocity | baseline and 10 minutes after induction
  The primary outcome was the end-diastolic velocity at 12 time points of anaesthesia induction among the three groups.

SECONDARY OUTCOMES:
pulsed-wave Doppler ultrasound | before leaving the PACU, up to 5 minutes
  other data related to pulsed-wave Doppler ultrasound and acquired during anaesthesia induction, before leaving the PACU and during inspiratory cough
intraoperative consumption of phenylephrine | through study completion, an average of 3 hours
  intraoperative consumption of phenylephrine

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, MD,PhD, Study Chair — Department of Anesthesiology
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided